CLINICAL TRIAL: NCT05404880
Title: Post-Market Clinical Follow-up Study of Edwards Lifesciences INSPIRIS RESILIA Aortic Valve in Chinese Population
Brief Title: INSPIRIS China PMCF Study
Acronym: INSPIRIS China
Status: Active, not recruiting | Type: Observational
Sponsor: Edwards Lifesciences (Industry)
Collaborators: Edwards (Shanghai) Lifesciences Medical Supplies Co., Ltd. (Industry); Rundo International Pharmaceutical Research & Development Co.,Ltd. (Industry); Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-09
Record Dates: First submitted 2022-05-31; First posted 2022-06-03 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- EDWARDS INSPIRIS RESILIA Aortic Valve: Subjects who were treated with the INSPIRIS RESILIA aortic heart valve.
  Interventions: Device: EDWARDS INSPIRIS RESILIA Aortic Valve

INTERVENTIONS:
Device: EDWARDS INSPIRIS RESILIA Aortic Valve — Surgical replacement of the aortic valve with the INSPIRIS RESILIA Aortic Valve.

SUMMARY:
The objective of this post-market trial is to evaluate long term safety and performance of the Edwards Lifesciences INSPIRIS RESILIA aortic valve in Chinese patients in a real-world clinical setting.

DETAILED DESCRIPTION:
The trial is a multi-center, prospective, single-arm study that will enroll up to 250 subjects. The study is being divided into 2 stages: Stage 1 is enrollment and 5 years of follow-up after implantation. Stage 2 is additional follow-up through 10 years upon authority's feedback if needed.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 18 years or older
2. Subjects requiring an elective replacement of their native or prosthetic aortic valve as indicated per the IFU
3. Subject is scheduled to undergo planned aortic valve replacement with or without concomitant coronary bypass surgery, with or without ascending aorta replacement
4. Provide signed informed consent prior to the study participation

Exclusion Criteria:

1. Valve implantation is contraindicated per the IFU
2. Requires planned multiple valve replacement/ repair
3. Has active endocarditis/myocarditis prior to the scheduled aortic replacement surgery
4. Estimated Life expectancy< 12 months
5. Current or recent participation (within 6 weeks prior to surgery) in another drug or device trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects requiring an elective replacement of their native or prosthetic aortic valve who have agreed to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Subject's Occurrence Rate of Study Valve Related Death | 5 Years
  The primary safety endpoint is the percentage of study valve related death which includes death caused by structural valve deterioration, nonstructural dysfunction, valve thrombosis, embolism, bleeding event, or operated valve endocarditis; death related to reintervention on the operated valve; or sudden, unexplained death.
Subject's Occurrence Rate of Structural Valve Deterioration | 5 Years
  The primary safety endpoint is the percentage of Structural Valve Deterioration which includes dysfunction or deterioration involving the operated valve (exclusive of infection or thrombosis), as determined by re-operation, autopsy, or clinical investigation.
Subject's Occurrence Rate of Re-operation on the Study Valve | 5 Years
  The primary safety endpoint is the reoperation rate on the study valve which is any operation that repairs, alters, or replaces the study valve, which occurs after the completion of the procedure and the transfer out of the procedure room.
Subject's Occurrence Rate of Major Bleeding | 5 Years
  The primary safety endpoint is the rate of major bleeding which is any episode of major internal or external bleeding that causes death, hospitalization, or permanent injury (e.g. Vision loss) or necessitates transfusion of 3 or more units of PRBC, pericardiocentesis, or exploration/reoperation for bleeding.
Subject's Occurrence Rate of Thromboembolic Events | 5 Years
  The primary safety endpoint is the rate of thromboembolic events which is an embolic event that occurs in absence of infection (endocarditis) starting from anesthesia time. Embolism may be manifested by a neurologic event (Stroke or Transient Ischemic Attack) or a non-cerebral embolic event.
Subject's Occurrence Rate of Stroke | 5 Years
  The primary safety endpoint is the rate of strokes which is a prolonged (>72 hours) or permanent neurologic deficit that is usually associated with abnormal results of magnetic resonance imaging or computed tomographic scans.
Subject's Occurrence Rate of Transient Ischemic Attack | 5 Years
  The primary safety endpoint is the rate of transient ischemic attacks which is characterized by fully reversible symptoms of short duration.
Subject's Occurrence Rate of Non-Cerebral Thromboembolism | 5 Years
  The primary safety endpoint is the rate of non-cerebral thromboembolism which is an embolus documented operatively, at autopsy, or clinically that produces signs or symptoms attributable to complete or partial obstruction of a peripheral artery (does not include deep vein thrombosis).

SECONDARY OUTCOMES:
Subject's Average Mean Gradient at 5 Years | 5 Years
  Hemodynamic performance - Mean gradients as evaluated by echocardiography
Subject's Average Peak Gradient at 5 Years | 5 Years
  Hemodynamic performance - Peak gradients as evaluated by echocardiography
Subject's Average Effective Orifice Area at 5 Years | 5 Years
  Hemodynamic performance - Effective Orifice Area evaluated by echocardiography
Subject's Average Effective Orifice Area Index at 5 Years | 5 Years
  Hemodynamic performance - Effective Orifice Area Index evaluated by echocardiography
Amount of Aortic Central Regurgitation in Subjects at 5 Years | 5 Years
  Hemodynamic performance - Aortic central regurgitation evaluated by echocardiography
Amount of Aortic Paravalvular Regurgitation in Subjects at 5 Years | 5 Years
  Hemodynamic performance - Aortic paravalvular regurgitation evaluated by echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Hansong Sun, Professor, Principal Investigator — Chinese Academy of Medical Sciences, Fuwai Hospital
Locations (13):
- China (13):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Beijing Anzhen Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Fuwai Hospital, CAMS & PUMC, Beijing, Beijing Municipality
  - Xiamen Cardiovascular Hospital Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Fuwai Hospital Chinese Academy of Medical Sciences, Shenzhen, Shenzhen, Guangdong
  - Henan Provincial Chest Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Fuwai Central China Cardiovascular Hospital, Zhengzhou, Henan
  - Nanjing First Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi
  - Sichuan Academy of Medical Sciences·Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Fuwai Yunnan Cardiovascular Hospital, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be available to other researchers.